CLINICAL TRIAL: NCT01554345
Title: Assessment of Preventive Effect of Vitamin E +Selenium on Acute Kidney Injury Through NGAL in Patients Undergoing Controlled Hypotension During Neurosurgery Operations
Brief Title: Effect of Vitamin E+Selenium on Kidney Function in Controlled Hypotension
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahed Hosein Khan, professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 89-04-30-11624
Record Dates: First submitted 2012-02-19; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: vitamin E +Selenium — vitamin E 400 IU once 8 hrs before operation selenium 150 mic once 8 hrs before operation

SUMMARY:
The purpose of this study is to determine whether Kidney injury happens in controlled hypotension during brain operations by using Neutrophil Gelatinase Associated Lipocalin ELISA Kit and if so, does VitaminE+Selenium prevent it

DETAILED DESCRIPTION:
NGAL(Neutrophil Gelatinase Associated Lipocalin) is a 25KD protein which bounds with Gelatinase in Neutrophil granules.It is also expressed in epithelial cells of kidney tubules.NGAL increases in ischemic and toxic injuries of kidney. During controlled hypotension in brain operations injury to the kidneys might occur . This study is designed to assess this possibility and evaluate the effect of VitaminE+Selenium on prevention of this problem

ELIGIBILITY:
Inclusion Criteria:

* All patients who are candidate for brain surgery under controlled hypotension

Exclusion Criteria:

* Positive history of renal disease
* Positive history of diabetes mellitus, CHF, HTN, Breast cancer, fever, leukocytosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
increased amount of urinary or serum NGAL after controlled hypotension | from 2 hours to 24 hours after controlled hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran university of medical sciences, Imam Khomeini Hospital, neurosurgery operation room and ward, Tehran, Tehran Province, Iran